CLINICAL TRIAL: NCT03103074
Title: Randomized Double Blind Placebo Controlled Pilot Study on Botulinum Toxin B as Treatment for Hidradenitis Suppurativa
Brief Title: Pilot Study on Botulinum Toxin B as Treatment for Hidradenitis Suppurativa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); Hidrosis Clinic, Stockholm, Sweden (Other)
Responsible Party: Principal Investigator, Øystein Grimstad, Md PhD, University Hospital of North Norway
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/149 (REK)
Record Dates: First submitted 2017-03-17; First posted 2017-04-06 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Hidradenitis Suppurativa
Keywords: botulinum toxin
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — rimabotulinumtoxinB; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: First treatment - one placebo and one active substance group Thereafter - all patients receive active substance
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Partcipant and investigator/outcomes assessor are blinded. Treatment will be given after randomization by a secondary investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum B Toxin (Experimental): Botulinum toxin B (Neurobloc(R)) 50 Units (U)/ml 0,05-0,1 ml/injection intradermally in a grid with 1- 1 1/2 cm between every injection in affected areas A maximum of 4000 U/patient/treatment Treatment every three months
  Interventions: Drug: Botulinum B Toxin
- Placebo (Placebo Comparator): Saline (NaCl 0,9%) 0,05-0,1 ml/injection intradermally in a grid With 1- 1 1/2 cm between every injection in affected areas Treatment in placebo group (n=10) only at first intervention
  Interventions: Other: Placebo Saline

INTERVENTIONS:
Drug: Botulinum B Toxin — Intradermal injections
  Other Names: Neurobloc
  Arms: Botulinum B Toxin
Other: Placebo Saline — Intradermal injections
  Other Names: Saline (NaCl 0,9%)
  Arms: Placebo

SUMMARY:
Randomized double blind placebo controlled pilot study/proof of concept-study to see if intradermal injection with Botulinum toxin B is an effective treatment of Hidradenitis suppurativa

DETAILED DESCRIPTION:
Twenty patients with hidradenitis suppurativa will be enrolled and randomised to treatment with either botulinum toxin B or placebo (saline) in affected areas.

Intervention and recording of data will be performed every three months. After three months, all patients will receive active substance. After six months, randomization will revealed. Patients with clinical improvement will be given the opportunity to continue treatment for additional six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active hidradenitis in the stage I-III according to Hurleys classification. Patients are referred to a dermatology out-patient clinic or patients already in an established treatment program, where there is indication for new or different treatment, or surgical intervention. Patients must have typical affection of the disease of either axillae, groins, and/or perigenital/perianal area

Exclusion Criteria:

* Patients in need of emergency medical or surgical treatment of hidradenitis will be excluded until the disease is in a quiet, controlled phase.

Pregnant or lactating, as well as patients with neurological disease such as myasthenia gravis or motor neuron disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
Patient reported improvement after invention with Botulinum toxin B | End point analysis 6 months
  Outcome measured by Dermatological Life Quality Index (DLQI)-scores

SECONDARY OUTCOMES:
Identification of clinical subgroups with best response to intervention as assessed by clinically scored measures | Interim analysis after 6 weeks- 3 months. End point analysis 6 months and sub group analysis 12 months
  Registration and analysis on investigator scored measures assessed by Hidradenitis suppurativa score (HiSCR) in relation to clinical phenotypes (location, Hurley stage)
Identify if covariates such as age, disease duration, smoking state, BMI and sweating influence patient reported improvement | Interim analysis after 6 weeks- 3 months. End point analysis 6 months and sub group analysis 12 months
  Covariate analysis on patient recorded DLQI in relation to pre-registered variables
Identification of clinical subgroups with best response to intervention as assessed by patient reported improvement | Interim analysis after 6 weeks- 3 months. End point analysis 6 months and sub group analysis 12 months
  Registration and analysis on patient recorded DLQI in relation to clinical phenotypes (location, Hurley stage)

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Grimstad, MD PhD, Principal Investigator — Consultant NEHR-HUD/Postdoc
Locations (1):
- University Hospital North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grimstad O, Kvammen BO, Swartling C. Botulinum Toxin Type B for Hidradenitis Suppurativa: A Randomised, Double-Blind, Placebo-Controlled Pilot Study. Am J Clin Dermatol. 2020 Oct;21(5):741-748. doi: 10.1007/s40257-020-00537-9. PMID 32761500